CLINICAL TRIAL: NCT02236585
Title: Does Patient-Controlled Epidural Bupivacaine-Fentanyl Offer Advantages Over Continuous Epidural Infusion After Uterine Arteries Embolization? A Controlled Prospective Study
Brief Title: Patient-Controlled Epidural Analgesia After Uterine Artery Embolization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UD-2015-16-P2Anesth; GPAnesth-2 (Other: Dammam University)
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Uterine Artery Embolization for Uterine Leiomyomata
Keywords: uterine artery embolization, epidural , patient-controlled analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient-controlled epidural analgesia (Active Comparator): Patient-controlled epidural analgesia
  Interventions: Procedure: Patient-controlled epidural analgesia
- Continuous epidural analgesia (Placebo Comparator): Continuous epidural analgesia
  Interventions: Procedure: Continuous epidural analgesia

INTERVENTIONS:
Procedure: Patient-controlled epidural analgesia — Patients will receive with patient controlled background infusion of 0.125% bupivacaine plus 2 μg/ml fentanyl that will be set between 4-6 ml/hour (to maintain visual analog scale (VAS) of ≥ 50 mm), intermittent bolus of 10 ml on demand by the women with lockout interval of 20 min with a four-hour maximum dose of 100 mL, irrespective of their age. The epidural infusions will be maintained for the first 24 postoperative hours
  Arms: Patient-controlled epidural analgesia
Procedure: Continuous epidural analgesia — Patients will receive continuous epidural infusion of 0.125% bupivacaine plus 2 μg/ml fentanyl at rate of 6-15 ml/hour (to maintain visual analog scale (VAS) of ≥ 50 mm).
  Arms: Continuous epidural analgesia

SUMMARY:
Uterine artery embolization (UAE) is commonly used to treat symptomatic uterine leiomyomata through induction of infarction and subsequent hyaline degeneration. This could be followed with variable severity of pain that lasts for several days after the procedure secondary to the resulted global uterine ischemia and fibroid infarction. Pain after UAE has been described as moderate to severe cramping increasing over the first 2 hours after UAE to reach plateaus for 5 to 8 hours before it rapidly decreases to a much lower level.1 The severity of pain after UAE seems unrelated to the uterine or fibroid size which makes the severity of pain is unpredictable.1

Pain management after UAE most often consists of a combination of a non-steroidal anti-inflammatory drugs, acetaminophen and an opioid. However severe pain following embolization of the uterine arteries may require large doses of parenteral opioids for relief with added unwanted effects.2

Additionally, patients received morphine intravenous patient-controlled analgesia (IV-PCA) after UAE needed considerable amounts of morphine (median [range] 24 mg [0-86 mg]) during the first 24 h after embolization.3 The addition of ketamine to IV-PCA failed to reduce morphine consumption for the first 24 hours after UAE. 2

Nowadays, the use of lumbar epidural anesthesia has been standardized as the anesthetic choice for uterine artery embolization as it improves patients satisfaction and reduces the severity of post-procedural pain.

Although some investigators suggest an epidural analgesia for pain control after UAE,4 the use of continuous lumbar epidural infusion of ropivacaine does not improve quality of pain management after UAE.5

Thus in an observational study included few patients, the investigators demonstrated considerable postoperative analgesia lasted for 24 hours after UAE with the combined use of patient-controlled thoracic epidural analgesia (PCEA) and rectal diclofenac.6 However, the catheterization of thoracic epidural space in such low-risk patients has many logistic issues.

Up to the best of our knowledge, there is no available comparative randomized clinical trial compares the use of continuous and patient-controlled lumbar epidural analgesia after UAE.

DETAILED DESCRIPTION:
The investigators hypothesize that the use of a patient-controlled lumbar epidural analgesia (PCEA) will reduce pain scores and improve patient's satisfaction after uterine artery embolization.

The present study is aiming to compare the efficacy of PCEA and continuous epidural infusion of bupivacaine 0.125% with fentanyl 2 µg/ml on the quality of postoperative analgesia after UAE. Furthermore, the investigators aim to study the correlations between the severity of pain after UAE and the number and size of uterine leiomyomata.

Following obtaining of the Local Ethics Committee approval and informed patient consent, sixty patients, aged 18years or older, undergoing routine elective UAE embolization for uterine leiomyomata under epidural anesthesia will be included in this prospective, randomized, controlled, double-blind, comparative study.

On the morning before embolization, the patients will be instructed in the use of the PCA pump and a VAS. The patients will be asked to rate their experienced pain using the VAS from 0 to 100 mm with 0 representing no pain and 100 representing the worst imaginable pain.

Prior to the procedure an 18 to 20 G intravenous access will be established. Patient monitors includes electrocardiograph, non-invasive blood pressure, peripheral oxygen saturation, and respiratory rate. All patients will be premedicated with iv midazolam 0.03 mg/kg.

A lumbar epidural catheter (22-G, B. Braun, Germany) will be placed in L2-4 position using loss of resistance to air and saline on the morning of the procedure. Aspiration and injection of a 3-mL test dose with 2% lidocaine will be used to exclude accidental intravascular or subarachnoid catheter position.

Anesthesia technique will be standardized for all women. A loading epidural dose of 20 ml of 0.25% bupivacaine with 2 μg/ml of fentanyl will be administered in divided 5 ml top-up doses. Epidural catheterization and anesthesia will be done by the attending anesthesiologists who will not be involved in the postoperative assessment of the patient and who is unaware of the patient's group.

Femoral artery will be cannulated with a 2.0 mm sheath of the embolization catheters and UAE will be performed by the same expert interventional radiologist with use of 355-500 μm polyvinyl alcohol particles (Boston Scientific and Cordis, Natick, MA, USA) suspended in 10 ml of iodixanol 270 mg I/ml (Visipaque; Nycomed Amersham, London, UK) mixed with 20 ml of isotonic saline. Embolization will be continued until cessation of UAE blood flow occurs.

After the completion of the procedure and decannulation of the femoral artery, the patients will be randomly allocated into two groups using computer generated randomization codes included in sealed opaque envelopes

According to our adopted protocol, all patients will receive iv infusion of paracetamol 1 g every 6 hours and lornoxicam 8 mg every 12 hours. if patients reached a VAS of ≥ 70 mm despite achieving the maximum preset hourly infusion rates (i.e. 15 ml/hour and 6 ml/hour in the CEA and PCEA groups, respectively), the protocol allows the attending anesthesiologist, who will not be involved in collection of patient data, to unlock the pump temporarily to administer epidural top-up doses of 5 mL of 0.25% bupivacaine plus 2 μg/ml fentanyl every 10 min as required irrespective of the randomization code. If the top-up doses exceeds 25 ml without pain reduction of ≥ 20 mm, an iv bolus injection of 100 mg tramadol will be given.

At the same time, side effects like as nausea, vomiting, itching, hypotension and bradycardia will be assessed and recorded. Nausea and vomiting will be treated with iv granisetron 1 mg. Troublesome pruritus will be treated with chlorpromazine hydrochloride 25 mg im. The patients will be discharged from the hospital after a one-night stay in the hospital. After discharge, pain will be controlled with oral lornoxiacam and paracetamol-codeine.

Using retrospective data from our centre in women received the standard continuous epidural analgesia, a sample size of minimum 30 patients per group was calculated with a study power of 90% to detect a 20% statistically significant difference in the cumulative consumption of bupivacaine for 24-hours after UAE.

Data will be expressed as mean ± SD and analysed using Student 't' test, Mann-Whitney U test and chi square test where appropriate. Linear regression will be performed to define the correlation between the severity of pain as regarding the VAS and the number and size of uterine leiomyomata. P < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Routine elective uterine artery embolization
* uterine leiomyomata
* Epidural anesthesia

Exclusion Criteria:

* Cardiac disorder
* Pulmonary disorder
* Renal disorder
* Hepatic disorder
* Neuropsychiatric disorder
* Bleeding disorder
* Severe anatomical abnormalities of the vertebral column
* Contraindications to epidural analgesia
* Preoperative pain score > 70 mm
* Drug abuse
* Daily intake of analgesics
* Language or mental disorders

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative consumption of bupivacaine-fentanyl | 24 hours after procedure
  The cumulative consumption of bupivacaine-fentanyl for 24 hours after uterine artery embolization (UAE) will be recorded

SECONDARY OUTCOMES:
Quality of analgesia | every 2 hours intervals after uterine artery embolization
  The patients will be asked to rate their experienced pain using the postoperative pain visual analogue scale (VAS) from 0 to 100 mm with 0 representing no pain and 100 representing the worst imaginable pain, for both parietal and visceral pain during rest and upon coughing
Time for first request for rescue analgesia | 6 hours after surgery
  The time for first request for rescue analgesia (i.e. visual analog scale (VAS) ≥ 50)
Number of supplementary top-up doses required | 24 hours after surgery
  number of supplementary top-up doses required
Cumulated amounts of local anesthetic consumption | 24 hours after procedure
  Cumulated amounts of local anesthetic and tramadol consumption for 24-hours after UAE
Overall patient satisfaction | 24 hours after surgery
  using 100-mm visual analog scale (VAS) (0 very unsatisfied and 100 very satisfied)
Uterine leiomyomata | 24 hours before uterine artery embolization
  number and size of uterine leiomyomata

CONTACTS AND LOCATIONS:
Overall Officials: Bander F Aldhafery, MD, Principal Investigator — Chairman of Radiology Dept
Locations (2):
- Saudi Arabia (2):
  - King Fahd Hospital of Dammam University, Khobar, Eastern Province
  - King Fahd Hospital of the University, Khobar, Eastern Province